CLINICAL TRIAL: NCT03249831
Title: Pilot Study to Evaluate the Safety and Feasibility of Induction of Mixed Chimerism in Sickle Cell Disease Patients With COH-MC-17: a Non-Myeloablative, Conditioning Regimen and CD4+ T-cell-depleted Haploidentical Hematopoietic Transplant
Brief Title: A Blood Stem Cell Transplant for Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16453
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease; Sickle Cell Disorder; Hemoglobinopathies; Thalassemia; Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Sickle Cell Disorders; Hemoglobinopathies; Thalassemia; Anemia, Sickle Cell; Haploidentical Transplant; Nonmyeloablative Conditioning; CD4+ T cell; CD4+ T cell-depleted Hematopoietic Cell Transplant; Mixed Chimerism
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; Thalassemia | interventions — Cyclophosphamide; Pentostatin; Antilymphocyte Serum; thymoglobulin; Tacrolimus; Mycophenolic Acid; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- COH-MC-17 and immunosuppressants (Experimental): Participants receive COH-MC-17: a 21-day nonmyeloablative conditioning regimen (cyclophosphamide, pentostatin and rabbit anti-thymocyte globulin), followed by CD4+ T-cell-depleted Haploidentical Hematopoietic Transplant on Day 0.
  Immunosuppressants (tacrolimus and mycophenolate mofetil) given on Day -1 onwards until discontinuation post-transplant.
  The minimally manipulated transplant product is manufactured using the CliniMACS device.
  Interventions: Drug: Cyclophosphamide; Drug: Pentostatin; Drug: Rabbit anti-thymocyte globulin; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Biological: CD4+ T-cell-depleted Haploidentical Hematopoietic Transplant

INTERVENTIONS:
Drug: Cyclophosphamide — Orally daily
  Other Names: Cytoxan
Drug: Pentostatin — Intravenous
  Other Names: NIPENT
Drug: Rabbit anti-thymocyte globulin — Intravenous
  Other Names: Rabbit ATG; Thymoglobulin
Drug: Tacrolimus — Initially IV. If patient tolerates, convert to oral.
  Other Names: PROGRAF®
Drug: Mycophenolate mofetil — IV or oral
  Other Names: MMF; CellCept®; Myfortic
Biological: CD4+ T-cell-depleted Haploidentical Hematopoietic Transplant — Infusion
  Other Names: CD4+ T-cell depleted HaploHCT; CD4+ T-cell depleted hematopoietic progenitor cell (HPC) product

SUMMARY:
Blood stem cells can produce red blood cells (which carry oxygen), white blood cells of the immune system (which fight infections) and platelets (which help the blood clot).

Patients with sickle cell disease produce abnormal red blood cells. A blood stem cell transplant from a donor is a treatment option for patients with severe sickle cell disease. The donor can be healthy or have the sickle cell trait. The blood stem cell transplant will be given to the patient as an intravenous infusion (IV). The donor blood stem cells will then make normal red blood cells - as well as other types of blood cells - in the patient. When blood cells from two people co-exist in the patient, this is called mixed chimerism.

Most children are successfully treated with blood stem cells from a sibling (brother/sister) who completely shares their tissue type (full-matched donor). However, transplant is not an option for patients who (1) have serious medical problems, and/or (2) do not have a full-matched donor. Most patients will have a relative who shares half of their tissue type (e.g. parent, child, and brother/sister) and can be a donor (half-matched or haploidentical donor).

Adult patients with severe sickle cell disease were successfully treated with a half-matched transplant in a clinical study. Researchers would like to make half-matched transplant an option for more patients by (1) improving transplant success and (2) reducing transplanted-related complications.

This research transplant is being tested in this Pilot study for the first time. It is different from a standard transplant because:

1. Half-matched related donors will be used, and
2. A new combination of drugs (chemotherapy) that does not completely wipe out the bone marrow cells (non-myeloablative treatment) will be used to prepare the patient for transplant, and
3. Most of the donor CD4+ T cells (a type of immune cells) will be removed (depleted) before giving the blood stem cell transplant to the patient to improve transplant outcomes.

It is hoped that the research transplant:

1. Will reverse sickle cell disease and improve patient quality of life,
2. Will reduce side effects and help the patient recover faster from the transplant,
3. Help the patient keep the transplant longer and
4. Reduce serious transplant-related complications.

DETAILED DESCRIPTION:
This is a pilot study to determine the safety and feasibility of the COH-MC-17 regimen and ability of the regimen to induce a mixed chimeric status in severe sickle cell disease patients (hemoglobin SS or S-βº Thalassemia). The COH-MC-17 regimen consists of a non-myeloablative regimen (cyclophosphamide, pentostatin and rabbit-anti-thymocyte globulin (ATG)) followed by a CD4+ T-cell-depleted haploidentical hematopoietic cell transplant (HaploHCT).

ELIGIBILITY:
Inclusion:

1. Confirmed diagnosis of hemoglobin SS or S-βº Thalassemia sickle cell disease
2. Severe disease status as defined by presence of one or more of the following:

   1. Clinically significant neurologic event (stroke) or any neurological deficit lasting > 24 hours; or increased transcranial Doppler velocity (>200 m/s). A stroke is defined as a sudden neurologic change lasting more than 24 hours that is accompanied by cerebral magnetic resonance imaging (MRI) changes.
   2. History of ≥ 1 episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea).
   3. History of ≥ 2 severe vaso-occlusive pain crises (VOC) per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea). A severe VOC is defined as an episode of pain lasting more than 2 hours severe enough to require care at a medical facility. Note that priapism that lasts more than 2 hours and requires care at a medical facility is also considered a VOC.
   4. Osteonecrosis of ≥ 2 joints despite the institution of supportive care measures.
   5. Prior treatment with regular RBC transfusion therapy, defined as receiving ≥ 8 transfusions per year for > 1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome)
3. No HLA matched sibling or 10/10 matched unrelated donor
4. Related donor who:

   1. Is genotypically haploidentical on HLA-A, B, C and DRB1 loci AND
   2. Meets institutional criteria
5. Failed prior hydroxyurea therapy or have intolerance to hydroxyurea
6. Meets protocol specified organ function criteria
7. Women of childbearing potential or sexually active male: Agreement to use adequate contraception prior to study entry and 6 months post-transplant.

Exclusion Criteria

1. Prior stem cell transplant
2. Prior bone marrow transplant
3. Concurrent other investigational agents, chemotherapy, biological therapy or radiation therapy
4. Planned use of moderate and strong CYP3A4 inhibitors
5. Active infection
6. Major surgery within the last 30 days
7. Clinically significant liver fibrosis or cirrhosis if on chronic transfusion therapy > 6 months
8. Active malignancy (other than non-melanoma skin cancers)
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to any in the pre- or post-transplant regimen.
10. Women of childbearing potential: pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Toxicity per NCI-Common Terminology Criteria for Adverse Events version 4.0 | Day -22 to 2 years post-transplant
Unacceptable Toxicity at least possibly related to COH-MC-17 | Day -22 to Day +60 post-transplant
Mixed Chimerism defined as 30-90% donor cells | Day +60 post-transplant
Feasibility of producing an infusion ready CD4+ T-cell-depleted hematopoietic product | From apheresis to Day 0

SECONDARY OUTCOMES:
Adverse events of Grade 3 or higher | Up to 2 years post-transplant
Neutrophil count ≥ 500/mm3, time to recovery | Up to 2 years post-transplant
Platelet count ≥ 20,000/mm3, time to recovery | Up to 2 years post-transplant
Marrow failure | Up to 2 years post-transplant
Sickle cell disease related complications | Up to 2 years post-transplant
Non-relapse mortality | Up to 2 years post-transplant
Acute Graft versus Host Disease per 1994 Keystone Consensus Criteria | Day + 100 post-transplant
Chronic Graft versus Host Disease per 2014 National Institutes of Health Consensus Criteria | Day+ 180, + 1 year and +2 years post-transplant
Overall Survival | Up to 2 years post-transplant
Disease-Free Survival | Up to 2 years post-transplant
Event-Free Survival | Up to 2 years post-transplant
Disease Relapse | Up to 2 years post-transplant
Persistent post-immunosuppressant mixed chimerism | Up to 2 years post-transplant
  Between 5% and 95% donor chimerism at two years post- transplant, at least 6 months post- immunosuppressant
Persistent immunosuppressant -dependent mixed chimerism | +2 years post-transplant
  Between 5% and 95% donor chimerism at two years post- transplant and on immunosuppressant
Complete chimerism: >95% donor chimerism | +2 years post-transplant
Primary donor graft failure: Defined as < 5% donor chimerism by Day + 30 post- transplant | Day +30 post-transplant
Secondary donor graft failure: Defined as < 5% donor chimerism beyond Day +30 in patients with prior documentation of ≥ 5% donor cells by Day +30 | > Day + 30 up to 2 years post-transplant
Donor chimerism in blood | Day +30, Day +60, Day +100, Day+180, and +1 yr, +1.5 yr, +2yr post-transplant
Donor chimerism in bone marrow | Day + 100, Day + 180 and + 1 yr post-transplant
Percent HbS levels | Baseline, and then Day + 30, Day + 100, Day + 180, +1 yr, +1.5, +2yr post-transplant

OTHER OUTCOMES:
Ratio donor: recipient de novo thymic T cells | Up to 2 years post-transplant
Ratio donor: recipient FoxP3+ regulatory T cells | Up to 2 years post-transplant
Tolerance status of donor: recipient type T cells | Up to 2 years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rosenthal, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States